CLINICAL TRIAL: NCT06232928
Title: Early Versus Late Intermaxillary Elastics in Patients With Class II Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamU
Record Dates: First submitted 2023-10-30; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2021-03

CONDITIONS: Class II Malocclusion Division 1
Keywords: Class II malocclusion; early Class II elastics; conventional Class II elastics
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 1-Early group (Experimental): for the early group, patients were instructed to wear immediate light short Class II elastics from upper canines to lower second premolars for 24 hours except while eating and change the elastics every 12 hours.
  Interventions: Device: Early Class II elastics
- 2-Conventional group (Active Comparator): for the conventional group, conventional class II elastics were used on rigid stainless steel arch wires. patients were instructed to wear Class II elastics from upper canines to lower first molars for 24 hours except while eating and change the elastics every 12 hours.
  Interventions: Device: Conventional Class II elastics

INTERVENTIONS:
Device: Early Class II elastics — Participants were treated by a fixed orthodontic appliance with intermaxillary class II elastics to correct the class II malocclusion. patients were instructed to wear immediate light short Class II elastics from upper canines to lower second premolars for 24 hours except while eating and change the elastics every 12 hours.
  Arms: 1-Early group
Device: Conventional Class II elastics — patients were treated by a fixed orthodontic appliance with intermaxillary Class II elastics. patients were instructed to wear Class II elastics from upper canines to lower first molars for 24 hours except while eating and change the elastics every 12 hours after reaching to rigid stainless steel arch wires.
  Arms: 2-Conventional group

SUMMARY:
This clinical trial aimed to compare the effect of immediate light short Class II elastics versus conventional Class II elastics on the skeletal, dental and soft tissues in patients with Class II malocclusion.

Participants with class II malocclusion divided into 2 groups; early group wore immediate light short Class II elastics and conventional group wore conventional Class II elastics on rigid stainless steel arch wires.

DETAILED DESCRIPTION:
Instrument and procedures I. Diagnostic Procedures

1. Medical and dental history.
2. Comprehensive clinical examination. a. Extraoral examination. b. Intraoral examination. c. Functional examination.
3. Diagnostic records

   1. Photographs.
   2. Orthodontic study models.
   3. Radiographic records.
4. Treatment plan II. Interventions

<!-- -->

1. Placement of pre-adjusted edgewise fixed orthodontic appliance.
2. Disarticulation of occlusion by glass ionomer cement.
3. Selection of the proper elastics size.
4. Patient motivation and instructions.
5. Follow up. III. Methods of data collection.

<!-- -->

1. Cephalometric analysis.
2. Digital models analysis.
3. Smile analysis. IV. Statistical Analysis.

I. Diagnostic Procedures Detailed and comprehensive patient diagnosis was performed guided by the evaluation sheet used at the Department of Orthodontics, Faculty of Dentistry, Ain Shams University.

The diagnostic procedure included the following steps:

1. Medical and dental history Full history was obtained for each patient including patient's name, sex, age, chief complaint, medical and dental history.
2. Comprehensive clinical examination a. Extraoral examination Frontal examination Extraoral examination included the examination of the patient's facial type, symmetry, vertical facial proportions, and lip competence.

   Smile examination Comprehensive smile analysis was carried out including gingival display on smiling, smile arc, smile symmetry and width of buccal corridors. All the patients included in the study showed normal gingival display on smiling.

   Profile examination Examination of facial profile type, lip protrusion and nasolabial angle, lip competence and vertical facial proportions was carried on profile examination.

   b. Intraoral examination Full and detailed intraoral examination included number of teeth present in the oral cavity, oral hygiene, periodontal condition of all teeth, the presence of any caries, broken restorations, and missing teeth.

   Examining the malocclusion in all planes of space was performed as well. Molar relationship, canine relationships and overjet were determined. The overbite was assessed. The midlines were checked for any shift, and the posterior occlusion was checked to determine any presence of posterior crossbite. Arch form, palatal vault shape and depth were also clinically examined. Patients included into the study showed Class II canine relationship, increased overjet and proclined maxillary incisors.

   The functional occlusion was also examined, including discrepancy between the intercuspal position and the retruded contact position, the occlusion during lateral excursions was examined for working and non-working side contacts, and the occlusal guidance was checked during anterior excursions.

   c. Functional examination The breathing pattern of each patient was checked. Additionally, the tongue was examined to determine any abnormal posture or function. Mouth breathing patients were referred for consultation to check for patency of airway and remove any causes of respiratory obstruction prior to treatment.
3. Diagnostic records

   A full set of orthodontic records was taken for every patient as part of the routine procedure for the treatment of patients in the outpatient clinic of the Orthodontic Department, Ain Shams University, including:

   a. Photographs

   • Eight essential orthodontic extra-oral and intra-oral photographs For each case, a full set of extraoral and intraoral photographs were taken.

   • Standardized smile photographs Three standardized smile photographs frontal, 45 degrees, and profile photographs were taken. These photographs were taken immediately before starting to wear the elastics and after reaching Class I canines' relation and alignment and leveling. For standardization, several parameters were fixed during capturing of the photos; i. Camera

   • Settings

   • Position ii. Lens iii. Patient head orientation i. Camera A camera D5300 was used to capture the standardized photos. The same camera was used to capture all photos for standardization.

   • Settings The camera settings were fixed during capturing all the photos The manual mode was selected, and the settings were adjusted. The aperture was set at f/13, the shutter speed was set at 1/200. The flash compensation was set to -0.3 and the exposure compensation was set at -1. The built-in flash in the camera was used.
   * position The camera was set at a fixed distance from the patient by using 3 permanent marks on the floor. The tripod was always repositioned on these marks for a fixed distance between the camera and the patient.

   To standardize the camera position in space (horizontal and vertical axes), the camera was connected to the quick-releasing plate which mounts the camera on the tripod. The tripod had two spirit levels which were used to ensure that the mounted camera was not tilted in the horizontal or the vertical axes. The round spirit level was used to adjust the vertical axis of the camera. The horizontal spirit level was used to adjust the horizontal tilt of the camera. This was confirmed by ensuring that the air bubble was in the middle mark of the spirit level for every photo. The vertical level of the camera was raised till the focal point of the lens was at the same level of the patient's nasal tip.

   ii. Lens The focal length was set at 55 for all the photos. iii. Patient head orientation A fixed graduated gray background was placed behind the patients at a fixed distance from the patient and the camera was mounted on the tripod.

   Also, the graduated background was placed behind the patients. During the photography grids on the camera screen matched with grids of the graduated background. Once the patient sat on the chair. The patient's face mid-sagittal plane was parallel to lines drawn on the background and perpendicular to the floor. Finally, Patients were instructed to smile then the three photographs were taken. The choice of the post- elastics smiles photos was based on the selection of photos with equal lip elevation.

   b. Orthodontic study models Alginate impressions were taken for the upper and lower arches of each patient using suitable-sized perforated trays and alginate impression material mixed according to the manufacturer's instructions . Each impression was poured with improved orthodontic stone material . Orthodontic bases were established and trimmed for the study models. Then all models were scanned by a 3-shape R-750 scanner.

   c. Orthodontic Radiographic records
   * Lateral cephalometric radiographs A lateral cephalometric radiographic image was taken for each patient and was used to measure the anteroposterior and vertical skeletal, dental, and soft tissue relations.
   * Orthopantomogram radiograph An Orthopantomogram radiograph was taken and used to detect any dental or bone anomalies, and evaluate the general periodontal condition & bone level, stage of eruption & position of third molars.
4. Formulation of the problem list and treatment plan The information gathered from history, clinical examination, and diagnostic records was then used to formulate the problem list and eventually develop the treatment plan. If the treatment plan included non-extraction treatment with the use of pre-adjusted edgewise fixed orthodontic appliance and Class II elastics, the patient was included in the study.

Patients were then randomly allocated into the early or conventional groups and after having signed the informed consent, intervention procedures were then started.

II. Interventions

The procedures completed in this study were as follows:

Early group

In the early group, the pre-adjusted edgewise appliance was placed on both maxillary and mandibular arches either in the same visit or at least within the same week. Alignment and leveling were done using a standardized wire sequence. Immediate light short elastics were inserted from the first visit. The details are as follows:

1. Placement of Edgewise fixed orthodontic appliance Scaling, polishing, and oral hygiene instructions were given at least 1 week before bonding. Orthodontic brackets 0.018-inch slot size Roth prescription were then placed on upper and lower arch wires.
2. Disarticulation of occlusion by glass ionomer cement Glass ionomer cement was placed on the central fossa of the lower first molar bilaterally then the patient was instructed to close the mouth occluding on glass ionomer leaving a thin layer. This was then followed by removal of excess and finishing were done. Then Alignment and leveling were done using a standardized wire sequence.
3. Selection of the proper elastic size After bonding, disarticulation, and arch wires placement. The elastic size was chosen with the help of a force gauge. The elastics were selected based on the previously defined force range.

   Elastic was placed on the lower second premolar hook and stretched to the upper canine hook by force gauge while the patient occluded then the force level was checked if it was within the light force range (2-3.5 ounces) it would be selected.

   Patients were instructed on placement of the elastics using the elastic holder.
4. Patient motivation and instructions The importance of elastics was explained to patients to become motivated for regular elastic placement. Patients were instructed to change the elastics twice per day, 24 hours wear "remove it only while eating" and regularly mark the follow-up charts which were given to patients.
5. Follow up Patients were checked regularly during clinical visits every 4 weeks and arch wires were changed as usual. To encourage better patients' compliance, follow-up charts were regularly checked. Additionally, text messages were sent as reminders for the patients and they were asked to send photographs of their teeth with the elastics every two weeks.

Patients were followed up until the achievement of a Class I canine relationship and reaching to 0.016×0.022-inch arch wire stainless steel. Finally, the post-elastics records were taken as follows:

orthodontic study casts. standardized smile and intraoral photographs. cephalometric radiograph. All patients were instructed to wear settling elastics with Class II vector until finishing and removal of fixed appliance.

Conventional group

1. Placement of pre-adjusted edgewise fixed orthodontic appliance This procedure was done in a manner similar to the early group. Patients were followed up every 4 weeks and arch wires were changed as usual for alignment and leveling. Once the patient reached 0.016×0.022 stainless steel arch wires, the arch wires were left for at least 1 month. Then all records (orthodontic study models, extraoral standardized smile and intraoral photographs, and cephalometric radiograph) were taken before starting Class II elastics.

2. Disarticulation of occlusion by glass ionomer cement The occlusal disarticulation was done as previously described for the early group.

3. Selection of the proper elastic size For elastics size selection, the elastics were placed on the first molar hook and stretched to the upper canine hook level. Then the elastic size was selected if the measured force was within the medium force range (4-5 ounces).

4. Patient motivation and instructions 5. Follow up For the previous steps, all were done in a manner similar to the early group. The arch wires were not changed. The 0.016×0.022-inch stainless steel arch wires were left until Class I canines were achieved. After the achievement of Class I canine relation, the same procedures were done including post-elastic records taking and instructions for settling elastics wear.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition stage with fully erupted permanent teeth (excluding third molars).
* Patients with increased overjet.
* Patients with canine Class II malocclusion.
* Treatment plan involves the use of a pre-adjusted edgewise fixed orthodontic appliance with a non-extraction approach.

Exclusion Criteria:

* Patients with a gummy smile.
* Obvious periodontal disease and gingival recession.
* Vulnerable patients (orphans, subjects with mental disorders…. etc.).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
the change of the maxillary incisors inclination | from the beginning of the treatment till treatment was done about 15 months
  The primary outcome of this study was to compare the effect of early light short elastics versus conventional elastics on the inclination of upper incisors in patients with canine Class II malocclusion.
  the Sella-Nasion angle was measured " cephalometric radiographic analysis" in degrees.
  the angle representing the maxillary incisors inclination "S-N angle" was measured before and after treatment by both protocols, then the amount of changes were compared.

SECONDARY OUTCOMES:
the 3-dimensional effects of early light short Class II elastics versus conventional elastics on dental, skeletal, and soft tissues. | from the beginning of the treatment till treatment was done about 15 months
  • The evaluation of skeletal, dental, and soft tissues changes was done by customized cephalometric radiographic analysis including "linear and angular measurements". customized analysis was done by Dolphin software including Witts, Steiner, Mcnamara, Holdway, and Tweed. "degrees and mm" and digital model analysis "linear and angular measurements" through 3 shape software. "degrees and mm"
amount of gingival display during smile | from the beginning of the treatment till treatment was done about 15 months
  • The evaluation of Class II elastics on the change of amount of gingival display during the smile.
  the standardized smile photos were taken before and after treatment and "linear measurements representing the amount of gingival displays" in mm were done and the changes in gingival display were assessed and comparison between both groups was done.
treatment duration | from the beginning of the treatment till treatment was done about 15 months
  The assessment of treatment duration for both protocols was done. the number of total months were utilized to treat this malocclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, El-Abasaya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: no limit

DOCUMENTS (1):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT06232928/Prot_000.pdf